CLINICAL TRIAL: NCT05556642
Title: Relapsed and Refractory Hepatoblastoma: A Prospective Registry and Hepatic Tumors Research Consortium Initiative
Brief Title: Relapsed and Refractory Hepatoblastoma: A Prospective Registry and Liver Tumor Research Consortium Initiative
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: rrHBL Registry
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Relapsed Hepatoblastoma; Refractory Hepatoblastoma
MeSH Terms: conditions — Hepatoblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — The following biospecimens will be collected:
  1. Fresh/ Frozen/ FFPE Tissue (DNA and RNA extraction may occur)
  2. Optional biospecimens include:
     1. urine (stored)
     2. blood (DNA and RNA extraction may occur)
     3. saliva (stored and DNA extraction may occur)
     4. tissue for tumor modeling, drug testing, or other applicable cancer-related research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with relapsed/ refractory Hepatoblastoma
  Interventions: Other: Biospecimen collection

INTERVENTIONS:
Other: Biospecimen collection — Clinical information and biospecimens will be collected

SUMMARY:
There are limited data regarding the biology and treatment of relapsed/refractory hepatoblastoma (rrHBL). This project provides the infrastructure for acquisition of biological specimens, imaging, and correlative clinical data to facilitate biology studies and characterization of rrHBL. This registry will collect clinical, demographic, and pathological data, specimens (as available) and imaging from patients with rrHBL, prospectively. Cases are identified through:

1. Existing clinical and/or cancer registry databases
2. Referrals from clinicians, surgeons, or pathologists
3. Families initiating contact with Registry staff directly

DETAILED DESCRIPTION:
The following data/materials will be collected:

Clinical Data: Demographic data, date of diagnosis, pathology, radiological imaging data, signs and symptoms at diagnosis, molecular and biological data, staging details including sites of disease, detailed treatment data (e.g. types and dates of surgeries/interventional therapy (if any), medical/systemic therapy, radiotherapy), response to treatment (imaging and tumor markers), dates of progression, types of progression (local or metastatic), and follow-up data. The demographic and clinical data collected are abstracted and entered into an electronic data system secured by password protection. Collection of existing molecular and/or genomic data or analysis that has been performed will also be included.

Research Specimens:

Tissue (fresh/frozen/FFPE) from diagnosis and all subsequent timepoints where tissue was acquired (for example at each relapse and/or progression) will be requested for all enrolled patients and sent for central review to the study pathologist and stored in the rrHBL biorepository within the Cancer and Blood Disease Institute at Cincinnati Children's Hospital Medical Center. Future research testing may be conducted on this tissue.

Optional research specimens:

Pending consent specification of family/patient, and resources, specimens may be sent directly to collaborating laboratories to proceed with tumor modeling and drug testing, or other translational research with PI or designee via an Institutional Review Board approved project.

* Tumor Modeling, Drug Testing, or Other Applicable Cancer-Related Research (Fresh, frozen,): Prospectively collected or retained left-over tumor tissue samples and normal tissue (background liver) as available, for research purposes.
* Blood: prospectively collected at time of enrollment and at time of subsequent relapse
* Urine: prospectively collected at time of enrollment and at time of subsequent relapse
* Saliva: prospectively collected at time of enrollment or at one time point after enrollment

Registry clinical data will be correlated with biological/bioinformatic and genomic data. Data stored in the Registry may be used to provide statistical data for scientific presentations and for preparation of peer- reviewed manuscripts.

ELIGIBILITY:
Inclusion Criteria:

* All patients of any age with a suspected diagnosis (per treating oncologist/surgeon) or confirmed diagnosis of a rrHBL and all patients with Hepatocellular Malignant Neoplasm- Not Otherwise Specified (HCN-NOS) who are <6 years of age at the time of initial diagnosis
* To allow for tumor modelling to be performed with fresh tissue from these cases, patients with suspected rrHBL are eligible to enroll on study
* Unless the patient is deceased, all patients and/or one parent or legal guardian must provide written informed consent as well as HIPAA/release of information consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with relapsed or refractory Hepatoblastoma
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2032-09-01 (Estimated); Study Completion 2040-09-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of relapsed or refractory Hepatoblastoma | From enrollment until data analysis is complete - assessed up to 40 years
  To characterize rrHBL across all age groups with regards to demographics, presenting features, pathology, radiology, clinical course, treatments and response
Create biorepository of specimens | From enrollment until data analysis is complete - retained up to 40 years
  To create a biorepository of specimens from patients with rrHBL or suspected to have rrHBL to enhance molecular/biological investigations
Clinical data and biological data correlation | From enrollment until data analysis is complete - assessed up to 40 years
  To correlate registry clinical data with biological/bioinformatic data

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Somers, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Studies submitted from other researchers will be approved by the Hepatic Tumors Research Consortium Steering Committee (HTRC SC) and will have appropriate Institutional Review Board approvals/determinations received by the Registry staff.

REFERENCES:
- See also: Relapsed and Refractory Hepatoblastoma (rrHBL) Registry website — http://rrHBLRegistry.org
- See also: Relapsed and Refractory Hepatoblastoma (rrHBL) Registry website — http://rrhbl.org